CLINICAL TRIAL: NCT03331965
Title: A Randomized Controlled Trial of Metoclopramide Versus Placebo During Gastrojejunostomy Tube Placement for Facilitating Guidewire Advancement Through the Pylorus
Brief Title: Metoclopramide Versus Placebo for GJ Placement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00081892; Putman Seed Fund 2017-01 (Other: Duke Department of Radiology)
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Radiation Exposure; Enteral Nutrition
Keywords: Interventional Radiology; Metoclopramide; Gastrojejenostomy
MeSH Terms: interventions — Metoclopramide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metoclopramide (Experimental): A one-time dose of promotility agent (2 mL of Metoclopramide 5 MG/ML Injectable Solution in 8 mL saline IV) will be administered at the time of GJ placement. After administration of the pro-motility drug, the GJ placement procedure will be performed using conventional technique. An IR technologist observing the procedure will record the fluoroscopy time, air kerma, and chronological time will be recorded by an IR technologist at the following routine events during GJ tube placement procedures: 1) start of gastric insufflation, 2) needle access to the stomach, 3) wire intubation of the duodenum, 4) wire intubation of the jejunum, 5) and procedure completion.
  Interventions: Drug: Metoclopramide 5 MG/ML Injectable Solution
- Saline (Placebo Comparator): A one-time dose of a placebo (10 mL saline IV) will be administered at the time of GJ placement. After administration of the placebo, the GJ placement procedure will be performed using conventional technique. An IR technologist observing the procedure will record the fluoroscopy time, air kerma, and chronological time will be recorded by an IR technologist at the following routine events during GJ tube placement procedures: 1) start of gastric insufflation, 2) needle access to the stomach, 3) wire intubation of the duodenum, 4) wire intubation of the jejunum, 5) and procedure completion.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Metoclopramide 5 MG/ML Injectable Solution — A one-time dose of promotility agent (metoclopramide 10 mg in 10 mL saline IV) will be administered at the time of GJ placement.
  Other Names: Reglan
  Arms: Metoclopramide
Drug: Saline — A one-time dose of a placebo (10 mL saline IV) will be administered at the time of GJ placement.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The goal of this study is to determine whether use of promotility agents to stimulate gastric peristalsis can reduce fluoroscopy time and procedure time during gastrojejunostomy (GJ) tubes placement in interventional radiology (IR). The investigators hypothesize that increased gastric peristalsis will aid in advancing a guidewire through the pylorus, a time consuming and tedious step required during GJ tube placement. In order to maximize scientific rigor and clinical practice impact, the investigators aim to answer this question through a blinded, randomized, placebo controlled trial.

Specific Aim 1: To test the hypothesis that a single dose of IV metoclopramide immediately prior to GJ tube placement reduces the fluoroscopy time required to advance a guidewire through the pylorus.

Specific Aim 2: To determine whether a single dose of IV metoclopramide immediately prior to GJ tube placement reduces total procedure fluoroscopy time, air kerma and total procedure time.

Specific Aim 3: To assess the safety of a single dose of promotility agent prior to GJ tube placement by assessing rates of adverse events in the periprocedural period in patients receiving IV metoclopramide versus placebo.

DETAILED DESCRIPTION:
Gastrojejunostomy tube placement is a commonly performed procedure for providing nutritional support in patients unable to tolerate gastric feeds due to gastric outlet or duodenal obstruction or severe gastroesophageal reflux. When performed percutaneously, this procedure involves advancing a guidewire from the gastrostomy skin entry site through the pylorus. Based on data collected for quality improvement purposes the investigators have found that this step accounts for approximately one half the total fluoroscopy time and radiation dose during GJ tube placement and approximately one third of the total physician time in the procedure. Specifically, crossing the pylorus required on average 5.3 minutes of fluoroscopy time out of a total of 9.3 minutes for the entire procedure, and accounted for 92.2 mGy air kerma out of 201.7 mGy for the entire procedure. Furthermore, inability to advance a wire into the duodenum due to refractory pylorospasm is among the most common reasons for aborting GJ placement. Specifically, in approximately 1.5% of GJ placement procedures the pylorus cannot be crossed and a gastrostomy tube is placed instead. Only colonic interposition, in which GJ tube placement is not attempted, accounts for a larger fraction of failed procedures (3%). A variety of wire, catheter, and device related techniques have been described to facilitate wire intubation of the pylorus, but this remains a rate limiting step in the procedure. In order to reduce radiation doses to both the patient and interventional radiologist to levels that are as low as reasonably achievable and to maximize procedural success rates, adjunctive methods to aid in wire intubation of the pylorus are needed.

Previous meta-analyses of randomized controlled trials have found that a single dose of erythromycin or metoclopramide is effective at emptying the stomach of blood and improving visualization during endoscopy for upper gastrointestinal tract bleeding. Similarly, a previous randomized controlled trial demonstrated that a single dose of metoclopramide or domperidone increases the rate at which nasoenteric tubes spontaneously pass through the pylorus from 27 to 55%. Single dose metoclopramide is also indicated for reducing transit time during small bowel follow through examinations. Drug related adverse events in these studies were rare.

Although single dose promotility agents are established in the above described settings, they have not been studied for GJ tube placement. The investigators hypothesize that use of promotility agents may facilitate advancement of the guidewire through the duodenum and into the proximal jejunum during GJ tube placement by enhancing gastric peristalsis, pylorus relaxation, and small bowel motility. Single doses of promotility agents such as metoclopramide are inexpensive (approximately $1.02 per dose), easily administered at the time of the procedure, and have very favorable safety profiles. Therefore, promotility agents may represent a simple, effective, and readily feasible means of reducing radiation dose and procedure time during GJ tube placement, thus improving the safety and efficiency of this common IR procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* undergoing de novo GJ placement as part of their routine clinical care

Exclusion Criteria:

* Patient pregnant
* Contraindications to metoclopramide including:

  * allergic reaction
  * pheochromocytoma
  * QTc prolongation
  * history of seizure disorder
  * extrapyramidal symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Ronald, Principal Investigator — Medical Instructor, Vascular & Interventional Radiology
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Itkin M, DeLegge MH, Fang JC, McClave SA, Kundu S, d'Othee BJ, Martinez-Salazar GM, Sacks D, Swan TL, Towbin RB, Walker TG, Wojak JC, Zuckerman DA, Cardella JF; Society of Interventional Radiology; American Gastroenterological Association Institute; Canadian Interventional Radiological Association; Cardiovascular and Interventional Radiological Society of Europe. Multidisciplinary practical guidelines for gastrointestinal access for enteral nutrition and decompression from the Society of Interventional Radiology and American Gastroenterological Association (AGA) Institute, with endorsement by Canadian Interventional Radiological Association (CIRA) and Cardiovascular and Interventional Radiological Society of Europe (CIRSE). Gastroenterology. 2011 Aug;141(2):742-65. doi: 10.1053/j.gastro.2011.06.001. No abstract available. PMID 21820533
- [Background] Donnelly LF, Klosterman LA, Ball WS Jr, Bisset GS 3rd. Comparison of duodenal intubation techniques during conversion of gastrostomy to gastrojejunostomy tubes in children. AJR Am J Roentgenol. 1997 Dec;169(6):1633-4. doi: 10.2214/ajr.169.6.9393180. No abstract available.
- [Background] Bai Y, Guo JF, Li ZS. Meta-analysis: erythromycin before endoscopy for acute upper gastrointestinal bleeding. Aliment Pharmacol Ther. 2011 Jul;34(2):166-71. doi: 10.1111/j.1365-2036.2011.04708.x. Epub 2011 May 25. PMID 21615438
- [Background] Barkun AN, Bardou M, Martel M, Gralnek IM, Sung JJ. Prokinetics in acute upper GI bleeding: a meta-analysis. Gastrointest Endosc. 2010 Dec;72(6):1138-45. doi: 10.1016/j.gie.2010.08.011. PMID 20970794
- [Background] Hu B, Ye H, Sun C, Zhang Y, Lao Z, Wu F, Liu Z, Huang L, Qu C, Xian L, Wu H, Jiao Y, Liu J, Cai J, Chen W, Nie Z, Liu Z, Chen C. Metoclopramide or domperidone improves post-pyloric placement of spiral nasojejunal tubes in critically ill patients: a prospective, multicenter, open-label, randomized, controlled clinical trial. Crit Care. 2015 Feb 13;19(1):61. doi: 10.1186/s13054-015-0784-1. PMID 25880172
- [Background] Paul N, Rawlinson J, Keir M. The use of metoclopramide for the small bowel meal examination: pre-procedural versus peri-procedural oral administration. Br J Radiol. 1996 Dec;69(828):1130-3. doi: 10.1259/0007-1285-69-828-1130. PMID 9135468
- [Background] Lyon SM, Pascoe DM. Percutaneous gastrostomy and gastrojejunostomy. Semin Intervent Radiol. 2004 Sep;21(3):181-9. doi: 10.1055/s-2004-860876. PMID 21331127
- [Background] Pocock SJ. When (not) to stop a clinical trial for benefit. JAMA. 2005 Nov 2;294(17):2228-30. doi: 10.1001/jama.294.17.2228. No abstract available. PMID 16264167
- [Derived] DuRocher N, Smith TP, Gazda S, Olivas A, Whited K, Langston M, Jones D, Martin JG, Kim CY, Ronald J. Metoclopramide Reduces Fluoroscopy and Procedure Time during Gastrojejunostomy Tube Placement: A Placebo-Controlled Trial. J Vasc Interv Radiol. 2020 Jul;31(7):1143-1147. doi: 10.1016/j.jvir.2020.02.028. Epub 2020 May 23. PMID 32457012

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide | Saline
Started | 55 | 55
Completed | 45 | 51
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide | Saline | Total
Number analyzed (Participants) | 45 | 51 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (19.0) | 53.8 (17.7) | 55.3 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 38
  Male | 30 | 28 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 50 | 94
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 37 | 40 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Duodenal Intubation
Description: The fluoroscopy time required to advance a guidewire through the pylorus.
Time Frame: Up to 45 minutes.
Population: Participants who completed the study.
Measure: Mean (98% Confidence Interval); unit: Minutes
Arm/Group | Metoclopramide | Saline
Number analyzed (Participants) | 45 | 51
Minutes | 1.6 [0.3 to 10.1] | 4.1 [0.2 to 27.3]

2. Secondary Outcome: Total Procedure Fluoroscopy Time
Description: The total procedure fluoroscopy time.
Time Frame: Up to 1 hour.
Population: Participants who completed the study.
Measure: Mean (98% Confidence Interval); unit: Minutes
Arm/Group | Metoclopramide | Saline
Number analyzed (Participants) | 45 | 51
Minutes | 5.8 [1.5 to 16.2] | 8.8 [2.8 to 29.7]

3. Secondary Outcome: Total Procedure Air Kerma
Description: The total procedure Air Kerma (energy released in a unit mass of air) measured in milligray (mGy).
Time Frame: Up to 1 hour.
Population: Participants who completed the study.
Measure: Mean (96% Confidence Interval); unit: mGy
Arm/Group | Metoclopramide | Saline
Number analyzed (Participants) | 45 | 51
mGy | 91 [13 to 354] | 130 [24 to 525]

4. Secondary Outcome: Total Procedure Time
Description: The total procedure time.
Time Frame: Up to 1 hour.
Population: Participants who completed the study.
Measure: Mean (96% Confidence Interval); unit: Minutes
Arm/Group | Metoclopramide | Saline
Number analyzed (Participants) | 45 | 51
Minutes | 16.4 [8 to 51] | 19.9 [6 to 53]

5. Other Pre Specified Outcome: Number of Subjects Experiencing Adverse Effects in the Periprocedural Period
Description: To assess the safety of a single dose of promotility agent prior to GJ tube placement by assessing rates of adverse events in the periprocedural period in patients receiving IV metoclopramide versus placebo.
Time Frame: Up to 30 days after procedure.
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide | Saline
Number analyzed (Participants) | 45 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days from date of enrollment
Description: Collected on participants who completed the study.
Arm/Group | Metoclopramide | Saline
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/51
Other Adverse Events (participants affected / at risk) | 0/45 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metoclopramide (N=45) | Saline (N=51)
Hospitalization (Endocrine disorders) | 0 | 0
Inpatient Emergency Surgery (Gastrointestinal disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03331965/Prot_SAP_002.pdf